CLINICAL TRIAL: NCT00190112
Title: Change of Heart Rate Variability and Baroreflex Sensitivity After Ventral Cardiac Denervation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FEMH-E-940002
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2004-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

INTERVENTIONS:
Procedure: ventral cardiac denervation

SUMMARY:
Atrial fibrillation (Af) is the most common morbid event after open heart surgery. Its incidence ranges from 19% to 27%, as reported by the Society of Thoracic Surgeons database. Many groups have tried to understand and treat this difficult problem and have formulated different hypotheses to explain its origin. An imbalance of the autonomic nervous system after surgical intervention has been accepted as a major determinant for this morbidity. Ventral cardiac denervation is a fast and low-risk procedure. This intervention has shown significantly reduction of the incidence and severity of Af after routine coronary artery bypass surgery. This technique could be applied both on-pump or off-pump and used as an adjunctive procedure to achieve Af prophylaxis. However, the detailed mechanism remains unclear. Theoretically, heart receives its innervation from the autonomic nervous system (ANS) via the great vessels and pericardial attachment. The propensity and distribution of ANS nerve fibers are different in location. In this study, we would like to evaluate the ANS function after ventral cardiac denervation by using heart rate variability (HRV) and baroreflex (BRS) sensitivity. 30 patients proposed to have elective off-pump coronary artery bypass surgery are enrolled. After induction of anesthesia, the depth of anesthesia is controlled by inhalation agents and monitored by bispectral index. After the major cardiac operation, ventral cardiac denervation is performed by using electrocautery. The digital signals of heart rate and blood pressure are acquired before and after the surgical procedures under the same range of bispectral index (50~60). The paired HRV and BRS are analyzed. This will provide us more information to justify the procedure.

DETAILED DESCRIPTION:
Coronary artery bypass and ventral cardiac denervation:

Off-pump coronary artery bypass (OPCAB) is performed based on patient's coronary angiography. Following the completion of coronary anastomoses, ventral cardiac denervation is achieved by removing the nerves around the large vessels of the base of the heart that run from the right side of the superior vena cava and end at the level of the midportion of the anterior pulmonary artery. This was done by excising the fat pads that surround the superior vena cava, the aorta, and the anterior and right lateral aspects of the main pulmonary artery.

Hemodynamic study:

All patients underwent OPCAB have Swan-Ganz catheter in our institute. Cardiac output measurement is obtained by thermodilution method. Hemodynamic variables (systemic blood pressure, pulmonary artery pressure, central venous pressure, pulmonary capillary wedge pressure, systemic vascular resistance, and pulmonary vascular resistance, etc) are recorded during the measurement.

ECG and blood pressure monitoring system:

ECG and radial arterial blood pressure were recorded by an analog to digital converter system (National Instrument Inc.). The analog signals were digitized in a rate of 500Hz and were stored in a hard disk. The data were then analyzed by a program written with MATLAB language (version 5.2, MATHWORK Co.). QRS complexes were automatically classified and manually verified as normal sinus rhythm, arterial or ventricular premature beats, or noise by comparison of the adjacent QRS morphologic features. The N-N interval time series were then transferred to a personal computer and post-processed.

Data acquisitions:

Immediately after induction of anesthesia, the patient was intubated. Routine indwelling catheters, like CVP and SG catheter were inserted. Prior to skin incision, the depth of anesthesia was monitored by BIS system using bispectral index (60~70) and adjusted by inhalation agents. Digital ECG and BP signals were recorded for 15 min without any mechanical or pharmacological interference. After completion of surgical procedures, the data acquisition was repeated once again in the operation room under the same level of anesthesia.

Baroreflex sensitivity analysis:

The analysis of BRS was conducted by both the sequence method and the spectral (α-index) method. Sequence method: In brief, the beat-by-beat time series of systolic arterial blood pressure and ECG R-R intervals were scanned to identify sequences of over three consecutive beats in which the systolic blood pressure (SBP) and R-R intervals of the next beat changed concomitantly in increasing or decreasing sequence. Such beat-to-beat sequences were identified as baroreflex sequences. A linear regression was applied to the individual sequence and only r2 values >0.85 were accepted. The measure of each type of the integrated spontaneous BRS was obtained by averaging all accepted slopes of the same type during a 5-minute recording. Spectral (α-index) method: The α-index (α) was obtained by means of the simultaneous spectral analysis of the R-R intervals and the SBP variabilities, with the calculation being made from the square root of the ratio between the R-R intervals and the SBP variability in low frequency (LF) band (αLF, 0.04 to 0.15 Hz). The coherence between the R-R intervals and SBP was assessed by a cross-spectral analysis. The α-index was calculated only when the magnitude of squared coherence (K2) between the RR and the SBP signals exceed 0.5 in LF band.

Heart rate variability analysis:

The missing intervals of the raw N-N data were linearly interpolated and resampled at 4 Hz by the Ron-Berger method. Each 5-minute segment of N-N intervals was taken for HRV analysis. The time domain measurements of HRV included SDNN, r-MSSD. The frequency-domain measurements of HRV included LF and HF, which were calculated by Welch's averaged periodogram of the N-N intervals.

ELIGIBILITY:
Inclusion Criteria:

* Patients with normal sinus rhythm proposed to undergo coronary artery bypass surgery.

Exclusion Criteria:

* Patients with frequent atrial arrhythmia or paroxysmal Af were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Ming Chiu, M.D., Study Chair — Far Eastern Memorial Hospital